CLINICAL TRIAL: NCT04841317
Title: Implementing a Mobile Technology-Based System for Physician-Directed Remote Management of Hypertension: A Pilot Study
Brief Title: Mobile Technology for Blood Pressure Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Paul Wang, Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 59671; 20FRN35360178 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single-arm: Blood pressure intervention (Experimental): Participants will use a mobile technology system comprising of a remote home blood pressure monitoring cuff and a mobile application integrated with a clinician-facing component to view and manage remote blood pressures. Participants will use this for 12 weeks, with assessment of blood pressure outcomes and anonymous surveys regarding the technology at 12 weeks.
  Interventions: Combination Product: Mobile technology intervention

INTERVENTIONS:
Combination Product: Mobile technology intervention — Home blood pressure cuff used by patients twice a week, with blood pressures transmitted to providers remotely

SUMMARY:
The primary objective of this study is to assess the feasibility and effectiveness of a mobile-technology based system that integrates patient-facing and clinician-facing components to assist the management of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older with an established diagnosis of essential hypertension

Exclusion Criteria:

* Patients on more than 2 antihypertensives at time of enrollment
* Clinical diagnosis of secondary hypertension, that is, hypertension due to a secondary cause, including but not limited to the following:
* Renal artery stenosis
* Primary hyperaldosteronism
* Cushing syndrome
* Coarctation of the aorta
* Drug-induced hypertension
* Pheochromocytoma
* Obstructive sleep apnea
* Hospitalization for malignant hypertension or severe hypertension (including stroke, cardiac events, acute kidney injury) in the preceding 6 months
* Hospitalization for unstable angina or myocardial infarction in the preceding 6 months
* Prior diagnosis of heart failure or cardiomyopathy
* Stroke or transient ischemic attack within prior 6 months
* Prior organ transplantation
* Failure to obtain informed consent
* Pregnant or currently trying to become pregnant
* Patients who are enrolled in other research studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):e13-e115. doi: 10.1161/HYP.0000000000000065. Epub 2017 Nov 13. No abstract available. PMID 29133356
- [Background] Lewington S, Clarke R, Qizilbash N, Peto R, Collins R; Prospective Studies Collaboration. Age-specific relevance of usual blood pressure to vascular mortality: a meta-analysis of individual data for one million adults in 61 prospective studies. Lancet. 2002 Dec 14;360(9349):1903-13. doi: 10.1016/s0140-6736(02)11911-8. PMID 12493255
- [Background] Law MR, Morris JK, Wald NJ. Use of blood pressure lowering drugs in the prevention of cardiovascular disease: meta-analysis of 147 randomised trials in the context of expectations from prospective epidemiological studies. BMJ. 2009 May 19;338:b1665. doi: 10.1136/bmj.b1665. PMID 19454737
- [Background] Jaffe MG, Lee GA, Young JD, Sidney S, Go AS. Improved blood pressure control associated with a large-scale hypertension program. JAMA. 2013 Aug 21;310(7):699-705. doi: 10.1001/jama.2013.108769. PMID 23989679
- [Background] Logan AG, Irvine MJ, McIsaac WJ, Tisler A, Rossos PG, Easty A, Feig DS, Cafazzo JA. Effect of home blood pressure telemonitoring with self-care support on uncontrolled systolic hypertension in diabetics. Hypertension. 2012 Jul;60(1):51-7. doi: 10.1161/HYPERTENSIONAHA.111.188409. Epub 2012 May 21. PMID 22615116
- [Background] Logan AG, McIsaac WJ, Tisler A, Irvine MJ, Saunders A, Dunai A, Rizo CA, Feig DS, Hamill M, Trudel M, Cafazzo JA. Mobile phone-based remote patient monitoring system for management of hypertension in diabetic patients. Am J Hypertens. 2007 Sep;20(9):942-8. doi: 10.1016/j.amjhyper.2007.03.020. PMID 17765133
- [Background] Casey DE Jr, Thomas RJ, Bhalla V, Commodore-Mensah Y, Heidenreich PA, Kolte D, Muntner P, Smith SC Jr, Spertus JA, Windle JR, Wozniak GD, Ziaeian B. 2019 AHA/ACC Clinical Performance and Quality Measures for Adults With High Blood Pressure: A Report of the American College of Cardiology/American Heart Association Task Force on Performance Measures. J Am Coll Cardiol. 2019 Nov 26;74(21):2661-2706. doi: 10.1016/j.jacc.2019.10.001. No abstract available. PMID 31732293

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 participants signed informed consent; 30 were allocated to the study arm.
Groups:
- Blood Pressure Intervention: Participants use a home blood pressure monitoring cuff for 12 weeks, integrated with a mobile application to allow their clinician to remotely view and manage blood pressure.
Period: Overall Study
Arm/Group | Blood Pressure Intervention
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Blood Pressure Intervention
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.87 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 14
  Hispanic or Latino | 3
  Non-Hispanic Black | 2
  Non-Hispanic White | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 135 (10.01)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 86.2 (8.5)
Weight [Mean (Standard Deviation); unit: kg] | 84.82 (16.9)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.14 (5.09)
Chronic Kidney Disease (CKD) [Count of Participants; unit: Participants] | 1
Sodium [Mean (Standard Deviation); unit: mmol/L] | 141 (2)
Potassium [Mean (Standard Deviation); unit: mmol/L] | 4.3 (0.5)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.99 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Pressure
Description: Change in systolic and diastolic blood pressure (SBP and DBP).
Time Frame: Assessed at baseline and week 12
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Blood Pressure Intervention
Number analyzed (Participants) | 30
mmHg
  SBP | -14.5 [-19.2 to -9.8]
  DBP | -6.3 [-10.2 to -6.3]

2. Primary Outcome: Participant Survey
Description: A survey regarding usability and feedback about the intervention completed by participants. Questions 1 through 5 were rated on a scale of 1 (strongly disagree) to 7 (strongly agree); question 6 was rated on a scale of 1 (extremely confident) to 5 (extremely doubtful).
Time Frame: 12 weeks
Population: Participants who completed the survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blood Pressure Intervention
Number analyzed (Participants) | 11
score on a scale
  Q1: I consider myself to be technology savvy | 5 (2.1)
  Q2: I found the blood pressure cuff easy to use | 6.2 (0.75)
  Q3: I found it helpful to receive reminders to monitor my blood pressure | 4.9 (1.76)
  Q4: I made blood pressure measurement readings without difficulty | 6.2 (0.75)
  Q5: I found the app and blood pressure cuff convenient to manage my blood pressure | 5.2 (1.94)
  Q6: I am able to lower my blood pressure into a healthy range | 1.9 (1.14)

3. Primary Outcome: Physician Survey
Description: A survey regarding usability and feedback about the intervention completed by physicians. Physicians provided survey responses, but were not enrolled in the study. Questions 1, 2, and 3 were rated on a scale of 1 (strongly agree) to 7 (strongly disagree); question 4 was rated on a scale of 1 (extremely confident) to 5 (extremely doubtful); question 5 was rated on a scale of 1 (extremely pleased) to 7 (extremely displeased).
Time Frame: 12 weeks
Population: Participants who completed the survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blood Pressure Intervention
Number analyzed (Participants) | 1
score on a scale
  Q1: I consider myself to be technology savvy | 5 (NA) — Standard deviation not calculable for n of 1
  Q2: I found the dashboard helpful to view and manage patient blood pressure data | 5 (NA) — Standard deviation not calculable for n of 1
  Q3: Using this system blood pressure management is more efficient compared to usual care | 2 (NA) — Standard deviation not calculable for n of 1
  Q4: This system will be useful to control my patients' blood pressure to a healthy range | 2 (NA) — Standard deviation not calculable for n of 1
  Q5: How would you rate your overall satisfaction with the care provided by the Dashboard? | 5 (NA) — Standard deviation not calculable for n of 1

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Blood Pressure Intervention
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-07-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT04841317/Prot_001.pdf